CLINICAL TRIAL: NCT01711749
Title: Study of Bioequivalence Between Two Formulations of 20 mg Rosuvastatin Calcium Tablets, Administered Under Fasting to Healthy Volunteers of Both Genders, Being the Test Formulation Manufactured by Laboratorios Phoenix S.A.I.C.F/Argentina for GlaxoSmithKline Brasil Ltda. and the Reference Formulation (Crestor®) Commercialized by AstraZeneca do Brasil Ltda.
Brief Title: Rosuvastatin Calcium Bioequivalence Study - Fast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117120
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Active Comparator): 01 tablet, single dose, of Reference Product in period 1 and 01 tablet, single dose, of Test Product in period 2.
  Interventions: Drug: Crestor®; Drug: rosuvastatin calcium tablets
- Sequence 2 (Active Comparator): 01 tablet of Test Product in period 1, and 01 tablet, single dose, of Reference Product in period 2.
  Interventions: Drug: Crestor®; Drug: rosuvastatin calcium tablets

INTERVENTIONS:
Drug: Crestor® — Reference formulation is rosuvastatin calcium tablets, 20mg, currently commercialized by AstraZeneca do Brasil Ltda., under the trademark Crestor®
Drug: rosuvastatin calcium tablets — Test formulation is rosuvastatin calcium tablets, 20 mg, produced by Laboratorios Phoenix S.A.I.C.F/Argentina for GlaxoSmithKline Brasil Ltda.

SUMMARY:
This is an open-label, randomized, two treatment, two sequences, two periods crossover study, using a crossover 2x2 design, where each subject will be randomly assigned to reference or test formulation, in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
The objective of this study is to confirm if two formulations of rosuvastatin calcium 20 mg tablets are bioequivalent. Test formulation is rosuvastatin calcium 20 mg tablets - manufactured by Laboratorios Phoenix S.A.I.C.F/Argentina for GlaxoSmithKline Brazil Ltda., administration of one single-dose tablet. Reference formulation is rosuvastatin calcium 20 mg tablets (Crestor® 20 mg - AstraZeneca do Brasil Ltda.), administration of one single-dose tablet. Sixty-four healthy volunteers, of both genders, with age ranging from 18 and 50 years old, will receive test or reference formulation under fasting conditions, according to the randomization list. In each period, after administration of medication, blood samples are collected at the following times: 0:00 (prior to administration), 0:30, 1:00, 1:30, 2:00, 2:20, 2:40: 3:00, 3:20, 3:40, 4:00, 4:20, 4:40, 5:00, 5:30, 6:00, 7:00, 8:00, 10:00, 12:00, 24:00, 36:00, 48:00 and 72:00 hours. The comparative bioavailability of formulations is evaluated based on relevant pharmacokinetic parameters for statistical comparison. Such parameters are obtained directly from the determination of the drug active principle plasmatic concentration, based on the application of a non-compartmental pattern for the evaluation of these concentrations after the drug oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 18 to 50 years. Women can not be pregnant nor breastfeeding, and man and woman commit to use an efficient contraceptive method along the entire study period;
* Volunteers of Asian descent, due to differences in the pharmacokinetics of rosuvastatin in this group of people;
* Volunteers cholecystectomy;
* Female subjects of childbearing potential must not become pregnant during the study period, thus, should be sexually inactive through abstinence or use of contraceptive methods the failure rate <1%. Inactivity sexual abstinence should be consistent with the usual lifestyle of the subject. Periodic abstinence and withdrawal are not acceptable methods of contraception. Will be accepted as methods of contraception with failure rate less than 1%: oral contraceptives, either combined or progestogen alone, injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, Percutaneous contraceptive patches, intrauterine device (IUD) or intrauterine system (IUS ) that meets the failure rate <1%, double barrier method, partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject;
* Body mass index ≥ 18.5 or ≤ 29.9 kg/m²;
* Volunteers with good health conditions and without significant diseases at medical criterion, as per the Clinical History; Blood pressure, pulse and temperature are taken, Physical examination, ECG and complementary Lab examinations;
* The volunteer is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study;
* The volunteer must be able to understand nature and purpose of the study, including the risks and adverse effects and must show good intention to cooperate with the researcher and act according to the requirement of the entire trial, what is confirmed by the signature of an Informed Consent.

Exclusion Criteria:

* The volunteer has a known hypersensitivity to the drug being studied or to any chemically related compounds;
* History or existence of hepatic or GI diseases or any other condition that could interfere with the absorption, distribution, excretion or metabolism of the drug;
* Use of maintenance therapy with any drug but oral contraceptives;
* History of hepatic, renal, pulmonary, GI, neurological, hematological, psychiatric, cardiologic or allergic problem of any etiology that needs drug treatment or that the researcher considers it is clinically relevant;
* Current or chronic history of liver disease, or know hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstone);
* ECG findings, not recommended at the researcher's criterion to participate in the study;
* Results of complementary lab tests that are out of the values considered normal, according to this protocol guidelines, unless the researcher considers them non-clinically significant;
* Smoke abuse;
* Daily ingestion of more than five cups of coffee;
* History of alcohol or drug abuse;
* Use of regular medication along the two weeks that preceded the study commencement, or use of any other medication one week before the study commencement;
* Hospitalization for any reason up to 8 weeks before the first period of study;
* Treatment along three months before the treatment commencement of the study with any drug known because of its well-defined toxic potential to major organs;
* Participation in any pharmacokinetics study with collection of more than 300 mL of blood or ingestion of any experimental drug along six months before the treatment commencement of the study;
* Donation or loss of ≥ 450 mL of blood along the three months that preceded the study or donation of more than 1500 mL along the 12 months before the treatment commencement of the study;
* Positive result for βHCG in urine in female volunteer;
* A positive pre-study Hepatitis B surface antigen or positive Hepatites C antibody result within 3 months os screening;
* Female subjects not using a contraceptive method that meets the failure rate <1%;
* Any condition that prevents the participation in the study, according to the researcher's judgment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2013-03-13 (Actual); Study Completion 2013-03-13 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve 0-t (AUC) | Collections points from time 0 to 72 hours after the drug administration, evaluated in two periods.
  Drug concentration area under the curve versus time, calculated by trapezoidal methods of time 0 to time t, where t is the time related to the last drug concentration, experimentally determined above the Quantification Limit (QL).
Area Under the Curve 0-infinite (AUC) | Collections points from time 0 to 72 hours after the drug administration, evaluated in two periods.
  Drug concentration area under the curve versus time, (time 0) infinite-extrapolated, where AUC[0-infinite] = AUC[0-t] + Ct/k, where Ct is the last drug concentration, experimentally determined (above the quantification limit) in that k is the terminal phase clearance constant.
Half Life (T1/2) | Collections points from time 0 to 72 hours after the drug administration, evaluated in two periods.
  Half life is calculated as ln(2) / k
Maximum concentration (Cmax) | Collections points from time 0 to 72 hours after the drug administration, evaluated in two periods.
  Maximum concentration reached after drug administration
Time to Cmax (Tmax) | Collections points from time 0 to 72 hours after the drug administration, evaluated in two periods.
  Time to obtain the maximum concentration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bragança Paulista, São Paulo, Brazil

REFERENCES:
- See also: Results for study 117120 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117120?search=study&search_terms=117120#rs